CLINICAL TRIAL: NCT07109986
Title: An Open-Label Clinical Study of UB-VV410 in Subjects With Active Refractory Systemic Lupus Erythematosus or Lupus Nephritis
Brief Title: UB-VV410 in Subjects With Active Refractory Systemic Lupus Erythematosus or Lupus Nephritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UB-VV410CI002
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: UB-VV410; Lupus Nephritis; Systemic Lupus Erythematosus; IASO
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive UB-VV410
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UB-VV410（treatment group） (Experimental): Interventions: UB-VV410. Subjects will be consented and screened. Once subject eligibility is confirmed, the Investigator will be notified which dose the subject is assigned to receive. Eligible subjects will receive UB-VV410 at the assigned DL（dose level） on Study Day 1 (Day 1). Dose-limiting toxicities (DLTs) will be assessed for 28 days after UB-VV410 treatment. Safety will be assessed throughout the study. SLE/LN disease activity will be evaluated at approximately 1, 2, 3, 6, 9, 12, 18, and 24 months following UB VV410 administration.
  Interventions: Drug: UB-VV410

INTERVENTIONS:
Drug: UB-VV410 — Treatment with single dose of UB-VV410, intravenous injection at Day 1. Note: Subjects may receive retreatment with UB-VV410 if there are preliminary findings suggesting incomplete improvement and acceptable safety.

SUMMARY:
This is an open-label investigator-initiated trial (IIT) to assess the safety, efficacy, and PK（pharmacokinetic）/PD（pharmacodynamics ） of UB-VV410 in adult subjects with clinically active treatment-refractory SLE. The study population will include subjects with active LN (as defined by evidence of active inflammation on renal biopsy, referred to as the LN cohort) and subjects with active SLE without LN (ie, non-LN SLE, referred to as the non-LN cohort). It is expected that the safety profile of UB-VV410 will be similar in subjects with active LN and subjects with active non-LN SLE; thus, dose finding (DF) will be conducted in the 2 subpopulation cohorts combined. Dose expansion (DE) may be conducted separately in the LN and non-LN cohorts to characterize the preliminary efficacy of UB-VV410, as well as its safety and PK/PD, in each subpopulation.

The objective of this study is to determine the MTD（maximum tolerated dose）/MAD（maximum administered dose） and the recommended dose for subsequent studies of UB-VV410 in subjects with active LN and in subjects with active non-LN SLE. The DF portion will evaluate the safety profile of UB-VV410 administered at various DLs（dose levels）. The DE portion will further optimize the dose and define the safety profile and preliminary efficacy of UB VV410. The study will use the Bayesian optimal interval (BOIN) design to allocate subjects to various DLs to minimize exposure to subtherapeutic DLs while maintaining appropriate safety parameters. DF will be initiated with UB-VV410 administered IV and starting at DL1.

During DF, additional subjects may be backfilled at DLs found to be safe per the BOIN design and with promising activity. After DF of UB-VV410 has been completed, DE with up to 14 subjects per DL within each subpopulation cohort (eg, LN and non-LN cohorts) may be implemented at DLs less than or equal to the MTD/MAD and demonstrating efficacy to further characterize the toxicity, tolerability, PK/PD, and preliminary efficacy of UB-VV410 at the selected DLs. The DE portion will further characterize product safety and preliminary efficacy in order to optimize benefit/risk. The number of DLs for DE will be determined based on the safety, activity and PK/PD data observed from DF.

In addition, some subjects may receive retreatment with UB-VV410 if there are preliminary findings suggesting incomplete improvement and acceptable safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤65 at time of consent.
2. Provide voluntary written informed consent.
3. Documented medical records indicated SLE diagnosis or diagnosis of SLE according to the 2019 EULAR（European Alliance of Associations for Rheumatology）/ACR（American College of Rheumatology） classification criteria for SLE for at least 6 months.
4. Current or history of elevated anti-dsDNA（anti-double-stranded DNA ） and/or elevated anti-Smith antibody.
5. Alanine aminotransferase (ALT) ≤ 2.5 × ULN（upper limit of normal）, aspartate aminotransferase (AST) ≤ 2.5 × ULN, AND total bilirubin < 1.5 × ULN (or AST, ALT, and alkaline phosphatase < 5 × ULN, and total bilirubin ≤ 3 × ULN for subjects with Gilbert's syndrome
6. No ongoing coagulopathies requiring periodic replacement of clotting factors (eg, fresh frozen plasma, cryoprecipitate). Note: Subjects on a stable anticoagulant regimen > 6 months with activated partial thromboplastin time (APTT) ≤ 2.5 × ULN and international normalized ratio (INR) > 2 and < 3 are allowed on study.
7. No serious concomitant diseases or active/uncontrolled infections.
8. For LN-specific subjects: Active, biopsy-proven, proliferative LN with the classification of Class III or Class IV according to the 2018 revised ISN/RPS criteria. Note: Overlapping Class V is allowed.
9. For Non-LN SLE-specific subjects: SLEDAI-2K（Systemic Lupus Erythematosus Disease Activity Index 2000） score of ≥ 8 (including at least 4 points from non-laboratory assessments; ) and at least 2 BILAG（British Isles Lupus Assessment Group） B organ system scores, and/or at least 1 BILAG A organ system score, including, but not limited to, cardiac (peri- or myocarditis), respiratory (pleuritis or lung involvement), vascular, hematological and musculoskeletal.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. BILAG A for neuropsychiatric SLE.
3. Any acute, severe lupus-related flare that needs immediate treatment, such as acute pericarditis, catastrophic antiphospholipid syndrome, or acute CNS lupus (eg, psychosis, seizure).
4. Diagnosis of drug-induced SLE rather than idiopathic SLE.
5. Receiving hemodialysis or peritoneal dialysis.
6. History of previous bone marrow transplantation, gene therapy, adoptive cell transfer, or any kind of CAR T-cell therapy.
7. History of or active human immunodeficiency virus (HIV) infection.
8. Active hepatitis B (HepB) or hepatitis C (HepC). Note: Subjects with negative HepB virus DNA or a negative HepC virus RNA assay for viral load quantifications are permitted. Additionally, subjects who are positive for HepB surface antigen and/or anti-HepB core antibody with a negative HepB virus DNA are eligible.
9. Allergies to supportive medications required for CAR T-cell toxicity management (eg, tocilizumab).
10. Ongoing CNS diseases (eg, seizure disorder, tremor, history of cerebral vascular accident [CVA]/recurrent transient ischemic attack [TIA], cerebritis, substantial psychiatric disorder) that would preclude evaluation of immune effector cell-associated neurotoxicity syndrome (ICANS).
11. Serious and/or uncontrolled medical condition that, in the Investigator's judgment, would cause an unacceptable safety risk, interfere with study procedures or results, or compromise compliance with the protocol.
12. Major surgery within 12 weeks prior to administration of UB-VV410 or plans to undergo major surgery during the trial period and whom the Investigator considers to be at unacceptable risk.
13. Actively receiving treatment in other interventional clinical trials. Note: continued follow-up on previous trials is allowed for survivorship, but no further investigational agents or assessments will be allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-05-08 (Estimated); Study Completion 2030-07-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE（Common Terminology Criteria for Adverse Events） v5.0 | up to 24 months after UB-VV410 infusion
  Type, frequency, and severity of adverse events (AEs) and laboratory abnormalities
Maximum tolerated dose (MTD) or maximum administered dose (MAD) and the recommended dose for subsequent study of UB-VV410 | up to 24 months after UB-VV410 infusion
  MTD/MAD and the recommended dose for subsequent study of UB-VV410

SECONDARY OUTCOMES:
clinical response of SLE to UB-VV410 | up to 24 months after UB-VV410 infusion
  Systemic Lupus Erythematosus Responder Index 4 (SRI-4) response at specified timepoints
clinical response of SLE to UB-VV410 | up to 24 months after UB-VV410 infusion
  The proportion of subjects with low disease activity by Lupus Low Disease Activity State (LLDAS) at specified timepoints
clinical response of SLE to UB-VV410 | up to 24 months after UB-VV410 infusion
  The proportion of subjects in remission as measured by Definition of Remission in SLE (DORIS) remission criteria at specified timepoints
clinical response of LN to UB-VV410 | up to 24 months after UB-VV410 infusion
  Clinical responses at specified timepoints as evaluated by the proportions of subjects with LN who achieve complete renal response (CRR), primary efficacy renal response (PERR), and partial renal response (PRR)

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Mao, Doctor, Principal Investigator — Jiangsu Province Hospital, the First Afﬁliated Hospital of Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No